CLINICAL TRIAL: NCT05339425
Title: Construction of Chinese Osteoporotic Fracture Registration Network Platform and National Cooperative Network
Brief Title: Chinese Osteoporotic Fracture Registration Network Platform
Acronym: CORN
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Hospital (Other Government); Tianjin First Central Hospital (Other); Hebei Medical University Third Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Peking University Third Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Ruijin Hospital (Other); Affiliated Hospital of Nantong University (Other); Shanghai Changzheng Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Second Xiangya Hospital of Central South University (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); First Affiliated Hospital of Fujian Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Sichuan Province Orthopetic Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Daping Hospital, Army Medical Center of PLA (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Peking University Shenzhen Hospital (Other); General Hospital of Ningxia Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Beijing Jishuitan Hospital (Other); Zhejiang Hospital (Other); Shenzhen People's Hospital (Other); Xiangya Hospital of Central South University (Other); Beijing Friendship Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai East Hospital of Tongji University (Other); Zhongda Hospital (Other); First Affiliated Hospital of Jinan University (Other); Fujian Provincial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021YFC2501701
Record Dates: First submitted 2022-04-01; First posted 2022-04-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-03

CONDITIONS: Osteoporosis; Osteoporotic Fractures
Keywords: Database; Osteoporosis; Osteoporotic Fractures; Registration
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Osteoporotic fracture: No additional intervention will be administered.
  Interventions: Other: No additional intervention will be administered.

INTERVENTIONS:
Other: No additional intervention will be administered. — No additional intervention will be administered.

SUMMARY:
China has gradually entered an aging society, and the incidence of osteoporotic fractures is increasing rapidly. Although the harm of osteoporotic fracture is huge, its diagnostic rate in China is still low. China still lacks a national osteoporotic fracture registration system, which has been established in many countries. The purpose of this study is to establish a Chinese osteoporotic fracture registration network platform (CORN), which will be helpful for the long-term comprehensive management of osteoporotic fracture population in China. This platform will help to establish a large prospective clinical cohort database of osteoporotic fractures and high-risk population in China.

DETAILED DESCRIPTION:
Previous studies have shown that the screening, diagnosis and treatment rates of osteoporosis and osteoporotic fracture in China are still low. The goal of this study is to establish a nationwide multicenter osteoporotic fracture registration network platform, a national collaborative network, a large osteoporotic fracture research cohort and a national biological specimen bank in Chinese mainland.

About 100 hospitals covering 20 provinces, autonomous regions and municipalities will be selected as collaborators. Each collaborator is going to enroll at least 500 patients with osteoporotic fractures on average, and a total of 50000 subjects are planned to be enrolled in our study.

Subjects will be assessed as follows:

1. Questionnaire investigation: including demographic data, past medical history, reproductive history, menstrual/menopausal history, family history of osteoporosis and fractures, awareness of disease, diagnosis and treatment of osteoporotic fractures, etc.
2. Clinical features: including anthropometric data, clinical symptoms, physical examination, grip strength test, balance assessment, walking speed test, etc.
3. Fall risk assessment: assessed by the Short Physical Performance Battery (SPPB), the Falls Risk for Older People in the Community (FROP-Com) and Morse Fall Scale (MFS).
4. Imaging evaluation: including thoracolumbar spine x-ray, bone mineral density (BMD) measurement by dual-energy x-ray absorptiometry (DXA), Quantitative computed tomography (QCT) and high-resolution peripheral quantitative computed tomography (HR-pQCT).
5. Laboratory tests: including blood calcium and phosphorus levels, bone turnover markers, parathyroid hormone level, 25-hydroxyvitamin D, 24-hour urine calcium, etc.
6. Biological specimen collection: blood and urine specimens are plan to be obtained for further studies with informed consent.
7. Follow-ups: subjects will be followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria (any of the following):

* Patients with hip osteoporotic fracture.
* Patients with vertebral osteoporotic fracture.
* Patients with low T-score ( ≤ -2.5) and at least one risk factor (e.g., history of osteoporotic fractures in other sites, a parental history of hip fracture, age ≥ 65 years, BMI < 18.5kg/m2, current smoking).
* Patients with very low T-score (< -3.0).
* The ten year probability of fracture by FRAX: major osteoporosis fracture ≥20%, or hip fracture ≥3%.

Exclusion Criteria:

* Patients who are unwilling to participate in the trial, have poor compliance and do not sign informed consent.
* Patients judged as unqualified participants by clinicians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at high risk of fracture.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of patients enrolled in 3 years | 3 years
  The number of patients enrolled in Chinese Osteoporotic Fracture Registration Network Platform (CORN) in 3 years
Age distribution | 3 years
  Age distribution of enrolled patients
Sex ratio | 3 years
  Sex ratio of enrolled patients
Body Mass Index (BMI) of enrolled patients | 3 years
  Weight and height will be combined to report BMI in kg/m^2
Quality of life of enrolled patients | 3 years
  Quality of life will be assessed with a five-level EuroQol five-dimensional (EQ-5D-5L) questionnaire (Chinese version). Measurement results of EQ-5D-5L will be used to generate values with an EQ-5D-5L Value Set for China. And a higher value means a better QOL.
Fall risk assessment of enrolled patients | 3 years
  Fall risk will be assessed with Morse Fall Scale (Chinese version). The minimum value is 0, and the maximum value is 125. A higher value means a higher risk of fall.
Fracture risk Assessment of enrolled patients | 3 years
  Fracture risk will be assessed with Fracture Risk Assessment Tool (FRAX). And a higher value means a higher risk of fracture.
Bone turnover markers (BTMs) | 3 years
  BTMs of enrolled patients will be tested and analyzed.
Bone mineral density of enrolled patients | 3 years
  Bone mineral density (BMD) should be measured with dual energy X-ray absorptiometry (DXA).
Health record analysis | 3 years
  A comprehensive evaluation of patients' medical records, including symptoms, physical examination, treatments, etc.

SECONDARY OUTCOMES:
Follow-up rate after enrollment | Every year of the 3 years
  Follow-up rate after enrollment will be calculated
Usage rate of anti-osteoporosis drugs | Every year of the 3 years
  Usage rate of anti-osteoporosis drugs will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, MD, Study Chair — Peking Union Medical College Hospital
Locations (39):
- China (39):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Shijingshan Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Second Medical Center of The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital, Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fuzhou Second Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Lunjiao Hospital of Shunde Foshan, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - Guizhou Provincial Orthopedics Hospital, Guiyang, Guizhou
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's hospital of Changzhou, Changzhou, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Dalian Hospital of Chinese Traditional and Western Medicine, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Sichuan Province Orthopedic Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Fourth Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang